CLINICAL TRIAL: NCT04775901
Title: Application of Three-Dimensionally Printed Navigational Template in Percutaneous Transthoracic Lung Biopsy: A Prospective, Randomized, Controlled, Noninferiority Trial
Brief Title: Application of Three-Dimensionally Printed Navigational Template in Lung Biopsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Chang Chen, Prof. Dr., Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: L20-241
Record Dates: First submitted 2021-02-23; First posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Lung Neoplasms
Keywords: Biopsy, Needle; Printing, Three-Dimensional; Image-Guided Biopsy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT-guided lung biopsy (Other): Participants in this arm received conventional CT-guided percutaneous transthoracic lung biopsy.
  Interventions: Other: CT-guided lung biopsy
- Template-guided lung biopsy (Experimental): Three-dimensionally printed navigational template was designed based on the CT scan images acquired before the biopsy. Under the guidance of navigational template, percutaneous transthoracic lung biopsy was conducted.
  Interventions: Device: Template-guided lung biopsy

INTERVENTIONS:
Other: CT-guided lung biopsy — Percutaneous transthoracic lung biopsy was conducted stepwise under the real-time guidance of CT scan. This kind of modality served as an effective method for diagnosing peripheral lung lesions (all of the participants received fine-needle aspiration, some of them received coaxial needle biopsy as well, according to the pulmonologist's instruction).
  Arms: CT-guided lung biopsy
Device: Template-guided lung biopsy — A three-dimensional model consisting of participant's thoracic image information was initially reconstructed based on the CT scan data. Afterwards, a navigational template was customized, which accommodated well to the anatomical landmarks of the participant. The template was then printed by means of stereolithography from photopolymer material. Participants would receive navigational template-guided percutaneous transthoracic lung biopsy (all of the participants received fine-needle aspiration, some of them received coaxial needle biopsy as well, according to the pulmonologist's instruction).
  Arms: Template-guided lung biopsy

SUMMARY:
This is a prospective, randomized, controlled study to evaluate the diagnostic yield and safety of three-dimensionally printed navigational template in percutaneous transthoracic lung biopsy.

DETAILED DESCRIPTION:
The feasibility of three-dimensionally printed navigational template-guided percutaneous transthoracic fine-needle aspiration was validated by a phase I study. To further investigate the non-inferiority of navigational template-guided lung biopsy to conventional CT-guided modality in terms of diagnostic yield, this prospective, randomized, controlled, noninferiority trial was conducted.

ELIGIBILITY:
Ⅰ. Inclusion Criteria:

A. CT confirmed peripheral lung lesion;

B. Nodule size larger than or equal to 30 mm;

C. Scheduled for percutaneous transthoracic fine-needle aspiration;

D. Percutaneous transthoracic lung biopsy was conducted at supine or partially lateral decubitus;

E. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2;

F. Written informed consent provided.

Ⅱ. Exclusion Criteria:

A. Biopsy needle insertion route impeded by skeletal structures;

B. Lesion within 3 cm above diaphragmatic dome;

C. Insertion route longer than the biopsy needle;

D. Lung biopsy needed to be conducted at vertically lateral decubitus;

E. Any contraindication of percutaneous transthoracic lung biopsy;

F. Women who are pregnant or in the period of breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-11-25 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield of percutaneous transthoracic fine-needle aspiration | Three to four working days post-biopsy were needed to establish the diagnosis of the cytological specimens acquired by fine-needle aspiration.
  A percutaneous transthoracic fine-needle aspiration procedure was considered diagnostic if a malignant or specific benign diagnosis of the lesion was made. The ratio of diagnostic cases to all the participants who received the corresponding biopsy was considered as diagnostic yield.

SECONDARY OUTCOMES:
Diagnostic sensitivity of percutaneous transthoracic fine-needle aspiration | If an eventual diagnosis was attained by means of follow-up, a 12-month assessment was needed.
  All biopsy results that showed lung cancer were considered true positives (TP). For participants who had a nondiagnostic (intermediate or indeterminate) result from the first lung biopsy (fine-needle aspiration), subsequent diagnostic modalities including a re-biopsy, transbronchial needle aspiration or a 12-month follow-up was conducted to determine the final diagnosis. If any of these modalities demonstrated malignant, the case was considered a false negative (FN). Diagnostic sensitivity of the fine-needle aspiration procedure for lung cancer was defined as TP / (TP + FN).
Procedural duration | 15 mins post biopsy
  The length of procedural duration was measured from the time a patient lain on the examining bed of the CT scanner to the time the first CT scan post fine-needle biopsy was conducted.
Radiation exposure | 15 mins post biopsy
  The dosage of the radiation exposure the participant received during the process of fine-needle aspiration.
Complication rate | Real-time complication post biopsy indicates those recognized by the immediate CT scan, while delayed complication indicates those recognized by radiograph taken 4-6 hours post biopsy.
  Complication post fine-needle aspiration was evaluated by the first CT scan images post biopsy. Common complications include pneumothorax, pulmonary hemorrhage and hemoptysis. Complications needed further interventions were specially recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Chang Chen, MD, PhD, Principal Investigator — Shanghai Pulmonary Hospital, Tongji University School of Medicine
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang L, Li M, Li Z, Kedeer X, Wang L, Fan Z, Chen C. Three-dimensional printing of navigational template in localization of pulmonary nodule: A pilot study. J Thorac Cardiovasc Surg. 2017 Dec;154(6):2113-2119.e7. doi: 10.1016/j.jtcvs.2017.08.065. Epub 2017 Sep 1. PMID 29017792
- [Background] Zhang L, Wang L, Kadeer X, Zeyao L, Sun X, Sun W, She Y, Xie D, Li M, Zou L, Rocco G, Yang P, Chen C, Liu CC, Petersen RH, Ng CSH, Parrish S, Zhang YS, Giordano R, di Tommaso L; AME Thoracic Surgery Collaborative Group. Accuracy of a 3-Dimensionally Printed Navigational Template for Localizing Small Pulmonary Nodules: A Noninferiority Randomized Clinical Trial. JAMA Surg. 2019 Apr 1;154(4):295-303. doi: 10.1001/jamasurg.2018.4872. PMID 30586136